CLINICAL TRIAL: NCT04992663
Title: DELIVR: A Multicenter Randomised Controlled Trial Investigating the Effect of Virtual Reality on Labour Analgesia Use
Brief Title: Investigating the Effect of Virtual Reality on Labour Analgesia Use
Acronym: DELIVR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zuyderland Medisch Centrum (Other)
Collaborators: Diakonessenhuis, Utrecht (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: METCZ20210037
Record Dates: First submitted 2021-06-17; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Virtual Reality; Labor Pain; Labor Analgesia
Keywords: Virtual Reality; Analgesia; Labor Pain
MeSH Terms: conditions — Labor Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: Non-blinded, starting as single centre, randomised controlled trial (RCT). After implementation of the DELIVR trial in the Zuyderland MC, the study will be expanded as a multi centre trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (VR-group) (Experimental): The participants randomised into this group are offered the BirthVR intervention during Labour.
  The VR group receives a VR information moment during labour and the possibility to exercise with the VR glasses and they receive VR during labour from the moment they are in active labour and use VR as much as they prefer. After labour, participants of the VR-group receive a structured questionnaire in which tolerability, feasibility and satisfaction of VR use is evaluated and participants receive the WDEQ-B questionnaire and PROM and PREM (ICHOM; T3, T4, T5).
  As soon as VR does not serve as adequate pain relief during labour and a women requests additional pain medication this will be offered according to local protocol.
  Interventions: Device: PICO glasses and controller with BirthVR
- Care as usual group (No Intervention): Patients randomised to the care as usual group will be offered pain medication during labour according to the local protocol, and on maternal request only. Postpartum participants receive the WDEQ-B questionnaire and PROM and PREM (ICHOM; T3, T4, T5)

INTERVENTIONS:
Device: PICO glasses and controller with BirthVR — PICO glasses will be used for VR in the intervention group. BirthVR is a guided meditation VR application designed by qualitative research (VIREL study) performed by this study group.
  The BirthVR application contains the following components:
  * Information/introduction video (including a virtual reality tour through the labour ward of the Zuyderland MC)
  * Fase 1: Beach environment, guided meditation/breathing exercise (1 session: 25 minutes)
  * Fase 2: Underwater environment, guided meditation/breathing exercise (1 session: 25minutes)
  * Fase 3: Mountain environment, breathing technique exercise on demand by using the controller (1 session: 30 minutes)
  * Counseling video (cesarean section, epidural anesthesia)
  Arms: Intervention group (VR-group)

SUMMARY:
Childbirth is associated with labour pain and can be regarded as one of the most serious kinds of pain. Labour pain management methods include pharmacological and non-pharmacological methods. There is increasing evidence that virtual reality (VR) is effective in the reduction of pain. The implementation of alternative methods like VR to reduce labour pain can contribute to reduce the use of pharmacological pain management methods and associated side effects.

The objective of this study is to asses the effect of VR on the request for labour analgesia compared with standard care.

Secondary objectives are the effect of VR on; the referral rate from midwifery led first line care to second line obstetrical care, patient satisfaction of VR use, delivery expectancy and experience (WIDEQ-A and WIDEQ-B), patient reported outcome measures (PROMs) and patient reported experience measure (PREMs) as defined by international consortium for health outcome measures (ICHOM) and evaluate the social, economic, organizational and ethical issues of VR by using the health-technology assessment analysis (HTA).

Study design: The study concerns a non-blinded, single centre, randomised controlled trial Study population: Nulliparous and multiparous women with a singleton in cephalic presentation beyond 36+0 weeks' gestation and an intention for vaginal delivery.

The study population will be randomly assigned to the intervention group (VR-group) or the care as usual group. The intervention group will be exposed to an immersive guided relaxation VR experience (BirthVR) during labour. If a woman in the intervention group requires additional pharmacological pain relief, this will be offered according to the local protocol. The participants who are randomised to the standard care group receive labour pain analgesia on maternal request according to the local usual standard care.

DETAILED DESCRIPTION:
The study concerns a non-blinded single centre, randomised controlled trial (RCT).

Eligible patients will be randomised to either the VR group or standard care group. In addition to the standard care, the VR group receives a VR information moment during labour and the possibility to exercise with the VR glasses and they receive VR during labour from the moment they are in active labour and use VR as much as they prefer.

Patients randomised to the care as usual group will be offered pain medication during labour according to the local protocol, and on maternal request only.

Women in first line care will be informed and counseled by their own midwife during their 34 weeks checkup. Informed consent will be signed during their next checkup with 36 weeks. The patient will receive a study number together with their randomization group, during their next checkup the VR information video will be offered to women participating in the VR group. Women under hospital care during their pregnancy will be informed and counseled by their care giver in the Zuyderland MC during their 34 weeks checkup. At 36 weeks informed consent will be signed. Patients will then receive a study number together with their randomization group and during their next checkup the VR information video will be offered to women in the VR group.

Data will be collected during labour about VR. The following data will be collected; number of times VR is used during labour, number of minutes per VR session, dilatation and amount of contraction per 10 minutes when using VR for the first time and the way in which labour started.

After informed consent participating women will be randomly assigned the intervention group (VR group) or the care as usual group. Counseling will take place around 34 weeks of pregnancy. At 36 weeks of pregnancy randomization will be done by the data manager program. Stratified randomisation will be done to create equal groups concerning primiparous and multiparous women. After informed consent is obtained the women will be asked to fill in the ICHOM T2 questionnaire, a baseline questionnaire and the WDEQ-A questionnaire.

After labour, participants of the VR-group receive a structured questionnaire in which tolerability, feasibility and satisfaction of VR use is evaluated and participants receive the WDEQ-B questionnaire and PROM and PREM (ICHOM; T3, T4, T5). Postpartum participants of the care as usual group receive the WDEQ-B questionnaire and PROM and PREM (ICHOM; T3, T4, T5).

The study will be conducted in the Zuyderland Medical Center, location Heerlen and in first line midwifery practices (Verloskundig samenwerkings verband Zuyderland; VSV).

Subjects can withdraw from participating at any time for any reason without consequences. The investigator can decide tot withdraw a subject from the study for urgent medical reasons. After withdrawal of a participant, it is not possible to replace this participant with a new participant. After withdrawal of a participant, the patient is asked to agree using the data from the medical file.

The hypothesis is that BirthVR will result in a 15% decrease in the request for labour analgesia. Assuming a decrease of 15%, power of 80% and a type I error of 0.05, a total of 338 women must be included, of which 169 women in the BirthVR group and 169 women in the 'care-as-usual' group. Taking into account a loss to follow-up of 10%, 186 women will have to be included per study and a total of 372 women. It is expected to include 279 women in second line obstetrical care. The investigators expect to include 93 patients in first line midwifery care.

The data of both groups will be analysed using SPSS (version 27). A table with baseline characteristics will be compiled using the Mann-Whitney-U test. A Chi-square test will be used to answer our primary objective. If, after randomization, it appears that the groups still differ regarding certain (baseline) variables, possible confounders will be assessed using a multivariable linear regression analysis. A p-value of <0.05 will be considered statistically significant. Tolerability, feasibility and patient satisfaction of VR use will be assessed using the answers to the BirthVR questionnaire, WDEQ and ICHOM questionnaires, using mostly descriptive analyses. Missing values will be excluded or imputed depending on the number of missing values. If the missing data is less than 10% pairwise deletion will be used. If a participant is excluded or withdraws participation after being included but before even using VR, there will be a new participant included (1:1). A loss to follow-up of 10-20% will be corrected by a multiple imputation (SPSS). If the loss to follow-up is >20% the number of missing participants have to be included to protect the internal validity.

ELIGIBILITY:
Inclusion Criteria:

* Written and orally given informed consent
* 18 years and older
* Native Dutch speaker
* Singleton pregnancy
* Nulliparous or multiparous women
* cephalic presentation
* 36+0 weeks gestation
* Intention for a vaginal delivery
* Under care of Zuyderland hospital or one of the first line midwifery practices participating in the Verloskundig Samenwerkings Verband (VSV) Zuyderland

Exclusion Criteria:

* Chronic pain patients defined as 'persistent or recurrent pain lasting longer than 3 months. The pain is not due to an obstetrical problem.
* Chronic use of pain medication (opioids)
* Alcohol or drug abuse
* Known car sickness
* Epileptic insults in previous history
* Psychotically seizures in previous history
* Claustrophobic
* Visual impairment
* History of mental illness
* Patients in strict isolation (MSRA)
* Age <18 years
* Twin pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2021-06-17 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Change of request for pharmacological analgesia by women in labour | From the start of labour (contraction or spontaneous rupture of membranes) until start pushing (expulsion phase)
  Any pharmacological analgesia received during labour? Yes or no.

SECONDARY OUTCOMES:
The referral rate from midwifery led first line care to second line obstetrical care based on pharmacological analgesia request during labour | From the start of labour (contraction or spontaneous rupture of membranes) until start pushing (expulsion phase)
  Examine the referrals from midwifery led first line care to second line obstetrical care because of a wish for pain rmedication during labour.
Delivery expectancy and experience (WDEQ-A and WDEQ-B) | WDEQ-A (at 36week pregnancy), WDEQ-B (1-7 days post partum)
  The WDEQ is a 33-item, 6-point Likert scale questionnaire. Items refer to expectations and experiences before and after birth, each scoring from 0 to 6. Women have to answer while imagining how labour and delivery are going to be, and how they expect to feel. Items with positively formulated questions are reverse-scored. The sum score ranges from 0 to 165; the higher the score is, the greater the fear of childbirth.
Patient satisfaction of VR use and the application BirthVR (questionnaire) | 1-7 days post partum
  A patients' VR experience and satisfaction was examined using a post-intervention questionnaire.
  A short post intervention questionnaire (7 questions), intended to provide feedback about the experience and preference of the BirthVR application the patient used during labour. Ratings varied of very pleasant (+5) versus very unpleasant (0) and very much (+5) versus not at all (0).
  Theme's: General experience, reusing BirthVR, preference of environment, side effects.
Patient reported outcome measures (PROMs) as defined by ICHOM | AD 36weeks, 1-7 days post partum, 6 weeks post partum and 6 months post partum
  Outpatient clinic (AD 36 weeks) - Capture of patient reported outcomes according to timepoint T2 of the Dutch version of the ICHOM standard outcome set Pregnancy and Childbirth
  T1 = within 7 days postpartum
  - Capture of patient-reported outcomes according to timepoint T3 of the Dutch version of the ICHOM standard outcome set Pregnancy and Childbirth
  T2= 6 weeks postpartum - Capture of patient-reported outcomes according to timepoint T4 of the Dutch version of the ICHOM standard outcome set Pregnancy and Childbirth
  T3= 6 months postpartum
  - Capture of patient-reported outcomes according to timepoint T5 of the Dutch version of the ICHOM standard outcome set Pregnancy and Childbirth
Patient reported experience measure (PREMs) as defined by ICHOM | AD 36weeks, 1-7 days post partum, 6 weeks post partum and 6 months post partum
  Outpatient clinic (AD 36 weeks) - Capture of patient reported experiences according to timepoint T2 of the Dutch version of the ICHOM standard outcome set Pregnancy and Childbirth
  T1 = within 7 days postpartum
  - Capture of patient-reported experiences according to timepoint T3 of the Dutch version of the ICHOM standard outcome set Pregnancy and Childbirth
  T2= 6 weeks postpartum - Capture of patient-reported experiences according to timepoint T4 of the Dutch version of the ICHOM standard outcome set Pregnancy and Childbirth
  T3= 6 months postpartum
  - Capture of patient-reported experiences according to timepoint T5 of the Dutch version of the ICHOM standard outcome set Pregnancy and Childbirth

CONTACTS AND LOCATIONS:
Overall Officials: Martine Wassen, M.D., Principal Investigator — Zuyderland MC
Locations (1):
- Zuyderland MC, Heerlen, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No